CLINICAL TRIAL: NCT04371380
Title: A Phase 1, Open-Label Study to Evaluate the Pharmacokinetics and Tolerability of Cabotegravir and Rilpivirine Long-Acting Injections Following Intramuscular Administration in the Vastus Lateralis Muscle of Healthy Adult Participants
Brief Title: Pharmacokinetic Study of Cabotegravir and Rilpivirine Long-acting Intramuscular Injections in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: Janssen Pharmaceuticals (Industry); GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 208832
Expanded Access: NCT03462810 (Available)
Record Dates: First submitted 2020-04-28; First posted 2020-05-01 (Actual); Results first posted 2024-04-22 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
Keywords: cabotegravir; rilpivirine; HIV; Pharmacokinetics; intramuscular injection
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Rilpivirine; Injections

STUDY DESIGN:
Intervention Model Description: Eligible participants will receive orally, tablets of cabotegravir plus rilpivirine for 28 days. There will be 10 to 14 days wash out period followed by an IM injection of cabotegravir long-acting plus rilpivirine long-acting.
Masking Description: This is an open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OLI phase followed by Injection phase (Experimental): Participants will be administered cabotegravir at a dose of 30 mg plus rilpivirine dose of 25 mg once daily with meal on Day 1 to Day 28 in OLI phase. There will be 10 to 14 days wash out period after OLI. This will be followed by an injection phase, wherein participants will receive 600 mg cabotegravir long acting given as one 3 milliliter (mL) IM injection plus 900 mg rilpivirine long acting given as one 3 mL IM injection on Day 1.
  Interventions: Drug: Cabotegravir Tablets; Drug: Rilpivirine Tablets; Drug: Cabotegravir extended release suspension for injection (long-acting); Drug: Rilpivirine extended release suspension for injection (long-acting)

INTERVENTIONS:
Drug: Cabotegravir Tablets — Cabotegravir tablets will be white to almost white oval shaped film coated tablets with a unit dose of 30 mg and will be administered orally.
Drug: Rilpivirine Tablets — Rilpivirine tablets will be off-white, round, biconvex film coated tablets with a unit dose of 25 mg and will be administered orally.
Drug: Cabotegravir extended release suspension for injection (long-acting) — Cabotegravir long-acting will be a sterile white to slightly pink suspension containing 200 mg per mL of GSK1265744 as free acid for administration by intramuscular injection.
Drug: Rilpivirine extended release suspension for injection (long-acting) — Rilpivirine long-acting will be a sterile white suspension containing 300 mg per mL of rilpivirine as the free base for administration by intramuscular injection.

SUMMARY:
This is a phase 1, open label study in healthy participants to assess the pharmacokinetics of cabotegravir and rilpivirine in plasma following the administration of a single 600 milligram (mg) and a 900 mg intramuscular (IM) injection respectively, to separate vastus lateralis muscles on each leg. Cabotegravir is an integrase inhibitor being developed in combination with rilpivirine, a non-nucleoside reverse transcriptase inhibitor, for the treatment of human immunodeficiency virus (HIV). The objective is to evaluate pharmacokinetics, tolerability, and safety of cabotegravir long acting plus rilpivirine long acting administered concomitantly as two separate IM injections in the vastus lateralis muscle of adult healthy participants. The screening phase will be of 30 days, oral lead-in (OLI) phase of 28 days, there will be washout period of 10-14 days, followed by an injection phase and follow-up period will be up to 52-weeks. Approximately 15 adult healthy participants will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 18 to 50 years of age inclusive, at the time of signing the informed consent.
* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and cardiac monitoring.
* A participant with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range may be included only if the investigator in consultation with the medical monitor agree and document that the finding is unlikely to introduce additional risk and will not interfere with the study procedures. A single repeat of a procedure or laboratory parameter is allowed to determine eligibility.
* Participants who are negative on two consecutive tests for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2/COVID-19), performed at Screening and on Day -1 of admission to the Phase I unit, using an approved molecular test (polymerase chain reaction or antigen test).
* Body weight >=40 kilogram (Kg) and body mass index (BMI) within the range 18 to 35 kg per square meter (inclusive).
* Male or female. Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies. Male participants: Male participants are eligible to participate if they agree to the following during the intervention period and for at least 52 weeks after the last dose of study intervention; refrain from donating sperm plus either be abstinent from heterosexual or homosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent or must agree to use contraception/barrier as detailed; agree to use a male condom when having sexual intercourse with a woman of childbearing potential who is not currently pregnant, agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person. Female participants: a female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies; is not a woman of childbearing potential (WOCBP) or is a WOCBP and using a contraceptive method that is highly effective, with a failure rate of less than 1 percent (%,) during the intervention period and for atleast 52 weeks after the last dose of study intervention; the investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention; a WOCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 30 days of the first dose of study intervention, if a urine test cannot be confirmed as negative (e.g., an ambiguous result), a serum pregnancy test is required. In such cases, the participant must be excluded from participation if the serum pregnancy result is positive; the investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form.

Exclusion Criteria:

* Signs and symptoms which in the opinion of the investigator are suggestive of COVID-19 (example; fever, cough etc) within 14 days of inpatient admission
* Contact with known COVID-19 positive person/s in the 14 days prior to inpatient admission
* History or presence of/significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, neurological or psychiatric disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Abnormal blood pressure as determined by the investigator.
* Alanine transaminase (ALT) greater than 1.5 times upper limit of normal (ULN).
* Bilirubin greater than 1.5 times ULN (isolated bilirubin greater than 1.5 times ULN is acceptable if bilirubin is fractionated and direct bilirubin less than 35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* History of ongoing or clinically relevant seizure disorder within the previous 2 years, including participants who have required treatment for seizures within this time period. A prior history of seizure, with a seizure free period of at least 2 years, off anti-epileptics, may be considered for enrollment if the investigator believes the risk of seizure recurrence is low. All cases of prior seizure history should be discussed with the medical monitor prior to enrollment.
* QT interval corrected for heart rate (QTc) greater than 450 millisecond for male participants and greater than 470 milliseconds for female participants
* A participant, who has an underlying skin disease or disorder (i.e. infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria).
* A participant, who is considered to have insufficient musculature to allow safe administration of cabotegravir or rilpivirine in the opinion of the investigator will be excluded.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication to the completion of the follow-up visit unless in the opinion of the Investigator and ViiV medical monitor the medication will not interfere with the study procedures or compromise participant safety.
* Participation in the study would result in loss of blood or blood products in excess of 500 mililiter within 56 days.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Participant has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Presence of Hepatitis B surface antigen (HBsAg) at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention.
* Positive Hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention.
* Presence of the Hepatitis B core antibody (HBcAb) should also lead to exclusion from the study even if HBsAg is negative.
* Positive pre-study drug/alcohol screen
* Positive human immunodeficiency virus (HIV) antibody test
* Regular use of known drugs of abuse
* Regular alcohol consumption within 6 months prior to the study defined as an average weekly intake of >14 units for males or >7 units for females. One unit is equivalent to 8 grams of alcohol: a half-pint (~240 milliliter) of beer, 1 glass (125 milliliter) of wine or 1 (25 milliliter) measure of spirits.
* Urinary cotinine levels indicative of smoking or history or regular use of tobacco- or nicotine-containing products (e.g. nicotine patches or vaporizing devices) within 6 months prior to screening.
* Participant, who has a tattoo or other dermatological condition overlying the thigh region which may interfere with interpretation of injection site reactions.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2021-12-26 (Actual); Study Completion 2021-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Fifteen participants were enrolled in the study. All the 15 participants received treatment in Oral Lead-in Phase. 14 out of 15 participants received treatment in Injection Phase. All the 14 participants in Injection phase completed the follow up phase.
Groups:
- Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg: Participants received 30 mg of CAB tablets orally along with 25 mg of RPV tablets once daily with meal from day 1 to day 28 of oral lead-in (OLI) phase.
- Injection Phase - CAB 600mg + RPV 900mg: Participants received single intramuscular (IM) dose of 600 mg of CAB LA injection on left and 900 mg of RPV LA injection on right side of lateral thigh on day 1 of injection phase (IP).
- Follow-up Phase - CAB 600mg + RPV 900mg: Participant who received 600 mg of CAB LA 900 mg of RPV LA injection during injection phase returned for safety assessments and additional PK sampling post injection in follow-up phase.
Period: Oral Lead-in Phase (Up to Day 28)
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
Started | 15 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Injection Phase (IP)-Day 1[IP] to Week 4
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
Started | 0 | 14 (14 participants transferred from OLI to injection phase) | 0
Completed | 0 | 14 | 0
Not Completed | 0 | 0 | 0
Period: Follow-up Phase (Week 4 to Week 52)
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
Started | 0 | 0 | 14 (14 participants transferred from injection phase to follow-up phase)
Completed | 0 | 0 | 14
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled population included participants who signed the informed consent form and received at least 1 dose of study drug.
Groups:
- All Enrolled Participants: Participants who signed the informed consent form and received at least 1 dose of study drug.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 34.3 (7.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1
  Black or African American | 7
  White | 7

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Concentration (Cmax) of Cabotegravir (CAB) Following Single IM Injection
Description: Blood samples were collected at indicated time points for pharmacokinetic (PK) analysis of CAB.
Time Frame: Day 1 (pre-dose, 1 hour, 2 hours) and one post-dose sample on day 2, day 4, day 5, day 8, day 10, day 15, day 17, day 22, day 28, week 8, week 12, week 24, week 36 and week 52
Population: Pharmacokinetic (PK) parameter population included all participants who underwent plasma PK sampling and have evaluable PK parameters estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter (ug/mL)
Groups:
- IM CAB 600 mg: Participants received single IM dose of 600 mg of CAB LA injection on left side of lateral thigh on day 1 of injection phase.
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 13
Microgram per milliliter (ug/mL) | 3.38 (66)

2. Primary Outcome: Cmax of Rilpivirine (RPV) Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Groups:
- IM RPV 900mg: Participants received a single IM dose of 900 mg of RPV LA injection on right side of lateral thigh on day 1 of injection phase.
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 14
nanogram per milliliter (ng/mL) | 93.5 (37.7)

3. Primary Outcome: Time of Cmax (Tmax) of CAB Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of CAB.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Median (Full Range); unit: Hour
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 13
Hour | 167 [166 to 1317]

4. Primary Outcome: Tmax of RPV Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Median (Full Range); unit: Hour
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 14
Hour | 131 [70.1 to 647]

5. Primary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to Time (AUC[0-t]) of CAB Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of CAB.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*microgram per milliliter (h*ug/mL)
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 13
Hour*microgram per milliliter (h*ug/mL) | 3612 (23)

6. Primary Outcome: AUC(0-t) of RPV Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 14
h*ng/mL | 143891 (33)

7. Primary Outcome: AUC From Time Zero Extrapolated to Infinity (AUC[0-infinity]) of CAB Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of CAB.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ug/mL
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 10
h*ug/mL | 3948 (21.5)

8. Primary Outcome: AUC(0-infinity) of RPV Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 11
h*ng/mL | 171953 (31.1)

9. Primary Outcome: Apparent Terminal Phase Half-life (t1/2) of CAB Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of CAB.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 10
Days | 21.4 (79.3)

10. Primary Outcome: t1/2 of RPV Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Days
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 11
Days | 137 (26.6)

11. Primary Outcome: Geometric Mean of Absorption Rate Constant (KALA) of CAB Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of CAB.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour (/h)
Arm/Group | IM CAB 600 mg
Number analyzed (Participants) | 10
Per hour (/h) | 0.00135 (79.3)

12. Primary Outcome: Geometric Mean of Absorption Rate Constant (KALA) of RPV Following Single IM Injection
Description: Blood samples were collected at indicated time points for PK analysis of RPV.
Time Frame: as for outcome 1
Population: PK parameter population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour (/h)
Arm/Group | IM RPV 900mg
Number analyzed (Participants) | 11
Per hour (/h) | 0.000211 (26.6)

13. Secondary Outcome: Number of Participants With Liver Related Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Time Frame: Up to 56 weeks
Population: Safety population included all participants who have taken at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
Number analyzed (Participants) | 15 | 14 | 14
Participants | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Liver Related Abnormalities
Description: Blood samples were collected to assess abnormalities related to liver.
Time Frame: Up to 56 weeks
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
Number analyzed (Participants) | 15 | 14 | 14
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All cause mortality, non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 56 weeks.
Description: Safety population included all participants who have taken at least 1 dose of study drug.
Arm/Group | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg | Injection Phase - CAB 600mg + RPV 900mg | Follow-up Phase - CAB 600mg + RPV 900mg
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 3/15 | 14/14 | 2/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral lead-in Phase - Cabotegravir (CAB) 30 Microgram (mg) + Rilpivirine (RPV) 25mg (N=15) | Injection Phase - CAB 600mg + RPV 900mg (N=14) | Follow-up Phase - CAB 600mg + RPV 900mg (N=14)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 3 (3) | 0 (0)
Feeling hot (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 4 (4) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 8 (8) | 0 (0)
Injection site induration (General disorders) | 0 (0) | 7 (7) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 14 (14) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 2 (2) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 6 (6) | 0 (0)
Injection site warmth (General disorders) | 0 (0) | 3 (3) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Scratch (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Abortion induced (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2020-08-13): https://cdn.clinicaltrials.gov/large-docs/80/NCT04371380/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT04371380/SAP_001.pdf